CLINICAL TRIAL: NCT04565639
Title: Hand Assistive Rehabilitation Orthotic Device Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberating Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 120190037
Record Dates: First submitted 2020-08-31; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Orthoses; Prostheses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental Power Hand Orthosis (Experimental): Participants will test the improved grip strength using the powered hand orthosis system.
  Interventions: Device: Powered Hand Orthosis
- Experimental Power Hand Orthosis - Tasks of Daily Living (Experimental): Participants will test the improved ability to perform tasks of daily living using the powered hand orthosis system.
  Interventions: Device: Powered Hand Orthosis

INTERVENTIONS:
Device: Powered Hand Orthosis — A prototype powered hand orthosis system designed to improve grip strength and improve ability to perform tasks of daily living.

SUMMARY:
The primary objective of this study is to evaluate pinch strength improvements and improvements in coordination and functional ability. Pinch strength measurements are made on subjects both with and without the device to evaluate the potential improvements. Also, coordination and functional testing is performed both with and without the device to compare performance under both conditions and evaluate potential improvement.

DETAILED DESCRIPTION:
This study tests the powered hand orthosis device on a small number of participants (up to 6). Research participants with neuromusculoskeletal impairments were recruited for the study and consented with an approved protocol. The study was conducted during 1 visit to LTI in Holliston, MA . The study consists of several assessments. Participants are surveyed for cognitive limitations and self-assessment of difficulties in completing tasks of daily living by completing surveys such as the Quickdash Questionnaire [1], the Mini-Mental State test [2], and the McGann Feedback form [3]. Pinch strength without and with the powered orthosis is evaluated. A selection of functional outcome measures are performed such as the Southampton Hand Assessment Procedure (SHAP) [4], the Nine-Hole Peg Test (NHP) [5], and the Box and Blocks Test (BBT) [6].

ELIGIBILITY:
Participants in this study must meet the following inclusion/exclusion criteria.

* Subjects diagnosed with one of these conditions- ALS, brachial plexus injuries, CVA hemiplegia, multiple sclerosis, muscular dystrophy, spinal cord injury, and traumatic brain injury
* Range of motion (ROM) and strength characterized by one of the following limitations:

  * Range of motion within functional limits (as determined by our OT consultant Deb Latour), but with limited pinch strength measured by a pinch meter of less than 2 pounds or manual muscle test grade of 3.
  * Limited range of motion of the wrist, thumb, index, and middle fingers as determined by a clinical occupational therapist
* Passive ROM within functional limits as determined by our OT consultant Deb Latour
* No tremors in the hand or arm
* Must be able to understand and follow up to 3 step directions for testing
* No other comorbidities that may affect their ability to use the device
* Modified Ashworth Scale assessment for spasticity of less than 2
* Greater than 18 years old
* Must be able to wear a powered hand orthosis device.
* Be able to make the required visit(s) to LTI for testing
* Mini-mental test [2] score greater than 18

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Sustained grip strength | 1 minute
  The sustained grip available for achieving activities of daily living that require a sustained grip

SECONDARY OUTCOMES:
Maximum Grip Strength | 10 seconds
  The maximum strength available for achieving activities of daily living
Accomplishing activities of daily living | 10 minutes
  Subjects were tested to accomplish a number of activities of daily living both with and without the device. Initial activities included the SHAP protocol and other activities that were identified by our occupational therapist consultant as relevant to the device.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Keough, Principal Investigator — Liberating Technologies, Inc.
Locations (1):
- Liberating Technologies, Inc, Holliston, Massachusetts, United States